CLINICAL TRIAL: NCT00811460
Title: A Double-blind, Crossover, Randomized, Placebo-controlled Study to Investigate the Effect of Two Different Doses of Taspoglutide IRF Administered as Continuous Subcutaneous Infusion on First- and Second-phase Insulin Secretion in Type 2 Diabetic Patients
Brief Title: A Study of Taspoglutide in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BP21844; 2008-003582-97
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — taspoglutide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Placebo; Drug: taspoglutide

INTERVENTIONS:
Drug: Placebo — sc for 4 days
Drug: taspoglutide — 300micrograms/day sc for 2 days
Drug: taspoglutide — 800 micrograms/day sc for 2 days

SUMMARY:
This crossover study will assess the effect of 2 doses of Taspoglutide on first- and second-phase insulin secretion in patients with type 2 diabetes. Patients will receive a continuous subcutaneous infusion of a)the Immediate Release Formulation (IRF)of Taspoglutide 300 micrograms/day for 2 days followed by Taspoglutide 800 micrograms/day for 2 days or b)saline placebo for 2+2 days. After a washout period of 10-15 days, patients will be crossed-over for further treatment;those receiving Taspoglutide in period 1 will receive placebo in period 2, and vice versa. On days 2 and 4 of each period, insulin secretion patterns will be assessed. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-65 years of age;
* type 2 diabetes mellitus;
* treated with diet and exercise alone, or in combination with stable metformin for at least 3 months prior to screening.

Exclusion Criteria:

* type 1 diabetes mellitus;
* type 2 diabetes duration of <3 months;
* treatment with any oral anti-hyperglycemic medication other than metformin monotherapy during last 3 months;
* treatment with insulin for >7 days within 6 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Incremental area under insulin concentration time curve relative to basal insulin concentration | First 10 minutes after glucose bolus

SECONDARY OUTCOMES:
Incremental area under insulin concentration time curve relative to basal insulin concentration | 10-120 minutes after glucose bolus
Adverse events, laboratory parameters | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Neuss, Germany